CLINICAL TRIAL: NCT02947308
Title: A Longitudinal Study Examining Three RDoC Constructs in Adolescents With Non-Suicidal Self-Injury
Brief Title: A Study Examining Adolescents With Non-Suicidal Self-Injury
Acronym: RDoC
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: PSYCH-2016-24795; 1R01MH107394-01A1 (NIH)
Record Dates: First submitted 2016-10-17; First posted 2016-10-27 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Self-Injurious Behavior; Deliberate Self-Harm
Keywords: Anxiety; Depression
MeSH Terms: conditions — Self-Injurious Behavior; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — De-identified saliva samples will be retained until the completion of the study. At the time of the completion, samples will be destroyed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adolescents with NSSI: 12-16 year old females who have a history of non-suicidal self-injury are included in this cohort. No interventions will be administered.
- Healthy Controls: 12-16 year old females with no history of non-suicidal self-injury are included in this cohort.

SUMMARY:
This study will examine longitudinal brain development in young adolescent girls with a history of Non-Suicidal Self-Injury (NSSI). Specifically, three constructs outlined by the the Research Domains Criteria (RDoC) will be examined through self-assessment, MRI, and a cognitive battery.

DETAILED DESCRIPTION:
This study is designed to study brain development in 12-14 year old females with a history of NSSI. Assessments will take place over the course of three years, with three visits per year - a total of nine visits.

The first visit will take place at the Ambulatory Research Center (ARC) at the Fairview Riverside hospital complex. This visit will include a number of questionnaires designed to gather information about the participant's physical and psychological health. Additionally, measures of intelligence quotient (IQ) and demographics will be assessed.

The second visit will again take place at the ARC. For this visit, participants will be asked to partake in the Trier Social Stress Test (TSST) in which they prepare a short, five-minute speech and deliver the speech to an audience with an additional task to follow. The TSST will be videotaped. Following the completion of this task, the participant will complete computer tests in order to measure things like attention and memory. During the second visit, five saliva samples will be collected to measure levels of the hormone Cortisol. The participant will need to collect additional saliva samples at home.

The third visit will take place at the University of Minnesota Center for Magnetic Resonance Research (CMRR) and will involve a brain MRI. Before the MRI the participant will be asked to provide a urine sample and complete a drug and pregnancy test. During the MRI, the participant will be asked to lie quietly in the scanner. The participant will do activities such as resting, listening to music, and playing games using a button box while in the scanner.

The participant will need to come in to complete these assessments twice more at one and two years following the completion of the first set of visits - a total of nine visits overall.

ELIGIBILITY:
Inclusion Criteria:

* 12-16 years old
* Female
* Has had first menstruation
* Willingness to have de-identified data shared with RDoC database

Inclusion Criteria - Adolescents with Non-Suicidal Self-Injury:

* Any history of self harm

Inclusion Criteria - Healthy Controls:

* No history of self harm

Exclusion Criteria:

* Male
* Pregnancy
* MRI Incompatibility
* IQ of less than 80
* Major Medical Illness
* Diagnosis of any of the following: Primary Psychotic Disorder, Bipolar Spectrum Disorder, Autism Spectrum Disorder, Current or Past Substance Use Disorder

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents with a history of NSSI will be recruited from community outlets such as flyers, as well as through social media (e.g., Facebook and Pandora). Additionally, these adolescents will be recruited through local clinicians who treat adolescent mood disorders. Healthy controls will be recruited through community outlets and social media.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2025-07-18 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Injurious Thoughts and Behaviors Interview (SITBI) | Baseline; 12 months; 24 months
  This scale will be used to assess NSSI frequency in the past month, past year, and lifetime; average age of onset; severity of injuries (number of injuries per episode, severity of tissue damage -- worst point and average), function (automatic versus social, negative versus positive) and other information.

SECONDARY OUTCOMES:
Change in Saliva Cortisol Levels | Baseline; 12 months; 24 months
  As a measure of stress response, cortisol levels will be measured after administration of the Trier Social Stress Test. This test is designed to measure HPA axis functioning in the context of an interpersonal threat. Intra- and inter-assay coefficients of variability will be calculated. Summary indexes including slope and area under the curve estimates of cortisol in response to threat and resting conditions will be used in subsequent analyses.
Change in Beck Scale for Suicidal Ideation (BSSI) | Baseline; 12 months; 24 months
  A 19-item interview, assesses current suicidal ideation, with ratings for active suicidal desire, specific suicide plans, and passive suicidal desire. If the adolescent is assessed to be at risk, a member of the research team will work with the family and the adolescent to develop a safety plan.
Change in Inventory of Depression and Anxiety Symptoms (IDAS) | Baseline; 12 months; 24 months
  The IDAS is a 54-item assessment that provides a score for 11 domains; we will focus on general depression, suicidality, traumatic intrusion, panic, and social anxiety.
Change in Rejection Sensitivity Questionnaire | Baseline; 12 months; 24 months
  This assessment measures predicted interpersonal sensitivity and difficulties.
Change in Personality Assessment Inventory, Adolescent Form (PAI-A) | Baseline; 12 months; 24 months
  A self-report personality indicator for adolescent populations based on 22 scales of psychological well-being.
Change in the Dot-Probe Task | Baseline; 12 months; 24 months
  A computerized assessment designed to assess attentional bias to threat, as well as provide a behavioral measure of "vigilance" to threat (reaction times for a spatial task influenced by the presence of emotion faces).
Change in Self Perception Profile for Adolescents | Baseline; 12 months; 24 months
  An assessment designed to evaluate and measure six self-concept domains: Scholastic Competence, Athletic Competence, Social Competence, Physical Appearance, and Behavioral Conduct and Global Self-Worth.
Change in Barratt Impulsiveness Scale (BIS) | Baseline; 12 months; 24 months
  This scale utilizes self-report measures of impulsiveness. It includes 30 items that are scored to yield six first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and three second-order factors (attentional, motor, and non-planning impulsiveness).
Change in UPPS-P | Baseline; 12 months; 24 months
  This measure will be used to determine "Negative Urgency", or the tendency of an individual to act impulsively while they are in a state of negative affect.
Change in the Emotional Go/NoGo task | Baseline; 12 months; 24 months
  This measure will be used to assess response inhibition in the context of negative emotion contexts.
Change in MRI Data | Baseline; 12 months; 24 months
  Cortical thickness, brain activation, and functional connectivity several key networks (fronto-striatal, fronto-limbic, and medial cortical network) will be measured using structural and functional MRI.
Change in Timeline Followback Method (TLFB) for NSSI | Baseline; 12 months; 24 months
  A calendar format measure to retrospectively collect behavioral data that was adapted from an instrument for alcohol use will be used measure NSSI episodes that had occurred in the year between each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Cullen, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - Ambulatory Research Center (ARC), Minneapolis, Minnesota
  - Center for Magnetic Resonance Research, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota